CLINICAL TRIAL: NCT04317573
Title: Effect on the Adherence to Glaucoma Eye Drops by Improving Patient Understanding and Using a Tele-reminder System: A Randomized Controlled Clinical Trial
Brief Title: Effect on the Adherence to Glaucoma Eye Drops by Improving Patient Understanding and Using a Tele-reminder System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Lai Yien, Senior Resident, National University Health System, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018/00289
Record Dates: First submitted 2020-03-16; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: A total of 59 patients were recruited for the study. Subjects were randomised into three groups: control (n=19), card only (n=20), card and tele-reminder (n=20) with an allocation ratio of 1:1:1. (Figure 1). Sample size was calculated based on similar drug adherence studies powered to detect a true difference in adherence rates with power at 80% and alpha at 5% - 20 patients per group were required.12,13
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalised card (Active Comparator): The personalised card was printed by the attending ophthalmologist for the patient via a web accessible software we have developed. The software allowed the reviewing physician to select the medications the patient was prescribed and auto-generate a personalised card that will be sent to the network printer. The card illustrated the patient's eye drop regime in a simple pictorial format using coloured pictures of the eye drop bottles and universally recognised symbols. It can be folded to a compact size of 11cm x 7.5cm to allow patients to carry around in their wallets. This card will be given to patients at the end of their consult and explanation will be provided by the attending physician who will manually tick in the corresponding boxes depending on the frequency of administration
  Interventions: Device: Personalised card
- Personalised card and telereminder (Active Comparator): Patients who were recruited into the group receiving tele-monitoring were contacted via text messages daily by a programmed software at the scheduled time of eye drop administration. They were required to acknowledge the reminder by replying a 'Yes' if they had administered the eyedrop and 'No' if they had not. A nil reply was taken as a 'No'.
  Interventions: Device: Personalised card
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Device: Personalised card — An individualised card containing the patient's eye drops regime was printed for the patient after his/consult with the physician to be brought home.
  Arms: Personalised card; Personalised card and telereminder

SUMMARY:
To determine the improvement in patient adherence to topical ocular hypotensive therapy by introducing a personalised illustrated medication reference chart and tele-reminder.

DETAILED DESCRIPTION:
This is a randomized controlled clinical trial study with patients recruited from the National University Hospital, Singapore who met eligibility criteria and agreed to participate in the study during their regularly scheduled outpatient visits. Written informed consent was obtained after the nature of the study had been fully explained to the patient. Recruitment took place from October 2018 to October 2019. The study received the local Institutional Review Board approval and all procedures are in accordance with the ethical standards as stated in the Helsinki Declaration.

A total of 59 patients were recruited for the study. Subjects were randomised into three groups: control (n=19), card only (n=20), card and tele-reminder (n=20) with an allocation ratio of 1:1:1. (Figure 1). Sample size was calculated based on similar drug adherence studies powered to detect a true difference in adherence rates with power at 80% and alpha at 5% - 20 patients per group were required.

The personalised card was printed by the attending ophthalmologist for the patient via a web accessible software we have developed. The software allowed the reviewing physician to select the medications the patient was prescribed and auto-generate a personalised card that will be sent to the network printer. The card illustrated the patient's eye drop regime in a simple pictorial format using coloured pictures of the eye drop bottles and universally recognised symbols. It can be folded to a compact size of 11cm x 7.5cm to allow patients to carry around in their wallets. This card will be given to patients at the end of their consult and explanation will be provided by the attending physician who will manually tick in the corresponding boxes depending on the frequency of administration.

Patients who were recruited into the group receiving tele-monitoring were contacted via text messages daily by a programmed software at the scheduled time of eye drop administration. They were required to acknowledge the reminder by replying a 'Yes' if they had administered the eyedrop and 'No' if they had not. A nil reply was taken as a 'No'.

Trained research assistants and a medical student administered the pre-implementation baseline adherence questionnaire in-person after informed consent was obtained. The questionnaire included questions on (i) demographics (ii) barriers to adherence and (iii) Morisky adherence scale. The demographic information included age, gender, length of time using glaucoma medications, number of glaucoma medications, educational level, whether they identify the medications by name or colour and who helps with the eye drop instillation. In the second section on barriers to adherence, participants were asked to use a visual analogue scale to rate the importance of 11 commonly cited reasons that make it "hard for patients to take glaucoma eye drops." The visual analog scale had 5 major hatch marks anchored between "strongly disagree" and "strongly agree." In the third section of the questionnaire, participants completed the Morisky Adherence Scale, a validated instrument for measuring self-reported adherence which was targeted for glaucoma medications in this study.

The interventions in both the card and tele-reminder groups were administered for a period of 6 weeks, following which a post-implementation adherence questionnaire was conducted via a telephone call by the same research assistants and medical student. The questionnaire included the same questions on the Morisky adherence scale as per the pre-implementation questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been treated for glaucoma for at least 3 months
* Using a total of three or more eye drops, at least two of which are ocular hypotensive
* A minimum visual acuity of 6/60 or better
* Aged 30 to 90 years old

Exclusion Criteria:

* Patients who just started on glaucoma treatment
* Patients who are on less than 3 eyedrops
* Patients with vision worse than 6/60

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2019-10-19 (Actual); Study Completion 2019-10-19 (Actual)

PRIMARY OUTCOMES:
Morisky Adherence Scale | 6 weeks
  Changes in mean adherence score based on Morisky Adherence Scale before and after intervention in participants from all 3 groups

CONTACTS AND LOCATIONS:
Overall Officials: Yien Lai, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- Yien Lai, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tham YC, Li X, Wong TY, Quigley HA, Aung T, Cheng CY. Global prevalence of glaucoma and projections of glaucoma burden through 2040: a systematic review and meta-analysis. Ophthalmology. 2014 Nov;121(11):2081-90. doi: 10.1016/j.ophtha.2014.05.013. Epub 2014 Jun 26. PMID 24974815
- [Result] Kass MA, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, Parrish RK 2nd, Wilson MR, Gordon MO. The Ocular Hypertension Treatment Study: a randomized trial determines that topical ocular hypotensive medication delays or prevents the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002 Jun;120(6):701-13; discussion 829-30. doi: 10.1001/archopht.120.6.701. PMID 12049574
- [Result] Heijl A, Leske MC, Bengtsson B, Hyman L, Bengtsson B, Hussein M; Early Manifest Glaucoma Trial Group. Reduction of intraocular pressure and glaucoma progression: results from the Early Manifest Glaucoma Trial. Arch Ophthalmol. 2002 Oct;120(10):1268-79. doi: 10.1001/archopht.120.10.1268. PMID 12365904
- [Result] Loon SC, Jin J, Jin Goh M. The relationship between quality of life and adherence to medication in glaucoma patients in Singapore. J Glaucoma. 2015 Jun-Jul;24(5):e36-42. doi: 10.1097/IJG.0000000000000007. PMID 24248002
- [Result] Olthoff CM, Schouten JS, van de Borne BW, Webers CA. Noncompliance with ocular hypotensive treatment in patients with glaucoma or ocular hypertension an evidence-based review. Ophthalmology. 2005 Jun;112(6):953-61. doi: 10.1016/j.ophtha.2004.12.035. PMID 15885795
- [Result] McDonald HP, Garg AX, Haynes RB. Interventions to enhance patient adherence to medication prescriptions: scientific review. JAMA. 2002 Dec 11;288(22):2868-79. doi: 10.1001/jama.288.22.2868. PMID 12472329